CLINICAL TRIAL: NCT02795962
Title: A Trial Comparing Transfer to the Closest Local Stroke Center vs. Direct Transfer to Endovascular Stroke Center of Acute Stroke Patients With Suspected Large Vessel Occlusion in the Catalan Territory.
Brief Title: Direct Transfer to an Endovascular Center Compared to Transfer to the Closest Stroke Center in Acute Stroke Patients With Suspected Large Vessel Occlusion
Acronym: RACECAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio Ictus Malaltia Vascular (Other)
Collaborators: Medtronic (Industry); Anagram-ESIC (Unknown); UPC (Unknown); BioClever 2005 S.L. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: RACECAT
Record Dates: First submitted 2016-06-01; First posted 2016-06-10 (Estimated); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Stroke
Keywords: Endovascular Procedures; Emergency Medical Services
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transfer to an Endovascular Center (Active Comparator): Acute stroke patients with suspected acute large vessel occlusion identified by EMS at first assistance on the field will be directly transferred to the nearest Endovascular Center bypassing the Local Stroke Center.
  Interventions: Other: Direct transfer to an Endovascular Center
- Transfer to the Local Stroke Center (No Intervention): Acute stroke patients with suspected acute large vessel occlusion identified by EMS at first assistance on the field will be transferred to the Local Stroke Center as done accordingly with the current stroke code protocol.

INTERVENTIONS:
Other: Direct transfer to an Endovascular Center — Cluster randomized controlled study: allocation to active or no intervention arm will be performed accordingly to a pre-established temporal sequence
  Arms: Transfer to an Endovascular Center

SUMMARY:
To evaluate the hypothesis that direct transfer to an Endovascular Stroke Center, compared to transfer to the closest Local Stroke Center, offers a better outcome in the distribution of the modified Rankin Scale scores at 90 days in acute ischemic stroke patients with clinically suspected Large Vessel Occlusion identified by Emergency Medical Services (EMS).

DETAILED DESCRIPTION:
Prospective, multicenter, cluster randomized controlled, usual care conditions, open, blinded-endpoint trial of acute stroke patients with suspected acute large vessel occlusion (LVO) identified by EMS at first assistance on the field, in which two strategies will be compared: transfer to the closest local stroke center (Local-SC) Vs. direct transfer to an endovascular stroke center (EVT-SC).

The RACE scale (Rapid Arterial oCclusion Evaluation) will be used as a prehospital screening tool to identify acute stroke patients with suspicion of LVO. Upon candidate identification, EMS will contact a stroke neurologist on call using a prehospital telestroke system who will confirm inclusion criteria and will allocate the subjects to a specific intervention according to a pre-established temporal sequence. Allocation will account for 3 strata: time band (two groups of 12 hours), territory (metropolitan versus provincial area) and week day (working versus weekend day).

Subjects will be followed up to 90 days post-randomization.

ELIGIBILITY:
Inclusion Criteria:

* Suspected LVO acute stroke patients identified by a RACE scale score >4 at the pre-hospital setting, that is evaluated by EMS professionals when attending patients, in non-stroke ready centers or primary health centers, previous to the transfer to a stroke center.
* Patients located in geographical areas in which the reference stroke center is a hospital not capable to offer endovascular treatment (Primary stroke Center or Telestroke Center).
* Estimated arrival time at an EVT-SC <7 hours from symptom onset. Symptom onset is defined as point in time the patient was last seen well (at baseline).
* No significant pre-stroke functional disability (modified Rankin scale 0 - 2)
* Age ≥18
* Deferred informed consent obtained from patient or acceptable patient surrogate (after the acute phase, as permission to use clinical data within a clinical registry)

Exclusion Criteria:

* Patients in a coma (NIHSS item of consciousness >1)
* Patients with unstable clinical status who require emergent life support care
* Serious, advanced, or terminal illness with anticipated life expectancy of less than 6 month.
* Suspected LVO acute stroke patients identified at the Emergency Department of a stroke center
* Subject participating in a study involving an investigational drug or device that would impact this study.
* Patients with a pre-existing neurological or psychiatric disease that would confound the neurological or functional evaluations. This excludes patients who are severely demented, require constant assistance in a nursing home type setting or who live at home but are not fully independent in activities of daily living (toileting, dressing, eating, cooking and preparing meals, etc.)
* Unlikely to be available for 90-day follow-up (e.g. no fixed home address, visitor from overseas).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1401 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
modified Rankin Scale score (shift analysis) | 90 days
  Modified Rankin Scale score in ischemic stroke patients as evaluated through a structured telephone-based interview performed by a central assessor who is blinded to group assignment.

SECONDARY OUTCOMES:
Mortality in all patients | 90 days
  Mortality in all patients included
Mortality in hemorrhagic stroke patients | 90 days
  Mortality in hemorrhagic stroke patients
Clinical deterioration requiring orotracheal intubation during transfers | 8 hours
  Orotracheal intubation during transfers
Clinical deterioration | 24 hours
  Clinical deterioration (≥4 points on the NIHSS)
Reperfusion therapies | 8 hours
  Proportion of patients receiving iv tPA and endovascular treatment within the first 8h from symptom onset
Time from symptom onset to reperfusion therapies | 8 hours
  Time from symptom onset to iv tPA administration (for patients treated with iv tPA) and to groin puncture (for patients treated with endovascular).
Subgroup analysis | 90 days
  Distribution of the modified Rankin Scale score at 90 days (shift analysis) in the following subgroups:
  * Ischemic / hemorrhagic
  * Patients eligible for iv t-PA vs. non iv t-PA eligible when attended by EMS (within time window considering transfer time to the nearest SC, no formal contraindications as recent major surgery or anticoagulation)
  * Patients treated with EVT
Clinical benefit of direct vs. local transfer accordingly with time and distance to the Endovascular Center | 90 days
  To analyze whether an inflection point exists with respect to time from onset to arrival at the Endovascular Center beyond which transfer to a Local-SC is beneficial or equivalent.
Dramatic early favorable response | 24 (-2/+12 hours)
  Dramatic early favorable response as determined by an NIHSS (National Institute of Health Stroke Scale) of 0-2 or NIHSS improvement ≥ 8 points in ischemic stroke and hemorrhagic stroke patients.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Ribó, PhD, Principal Investigator — Hospital Universitari Vall d'Hebrón, Barcelona, Spain; Sonia Abilleira, PhD, Principal Investigator — Pla Director Malaltia Vascular Cerebral. Agència de Qualitat i Avaluació Sanitàries de Catalunya (AQuAS); Natalia Pérez de la Ossa, PhD, Principal Investigator — Hospital Universitari Germans Trias i Pujol, Badalona, Spain
Locations (12):
- Spain (12):
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Bellvitge, Barcelona
  - Hospital Clínic, Barcelona
  - Hospital Mar, Barcelona
  - Hospital Moisés Broggi, Barcelona
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital Vall d'Hebrón, Barcelona
  - Hospital Josep Trueta, Girona
  - Hospital Arnau Vilanova, Lleida
  - Hospital Althaia, Manresa
  - Mutua Terrassa, Terrassa
  - Hospital Verge de la Cinta, Tortosa

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ramos-Pachon A, Rodriguez-Luna D, Marti-Fabregas J, Millan M, Bustamante A, Martinez-Sanchez M, Serena J, Terceno M, Vera-Caceres C, Camps-Renom P, Prats-Sanchez L, Rodriguez-Villatoro N, Cardona-Portela P, Urra X, Sola S, Del Mar Escudero M, Salvat-Plana M, Ribo M, Abilleira S, Perez de la Ossa N, Silva Y; RACECAT Trial Investigators. Effect of Bypassing the Closest Stroke Center in Patients with Intracerebral Hemorrhage: A Secondary Analysis of the RACECAT Randomized Clinical Trial. JAMA Neurol. 2023 Oct 1;80(10):1028-1036. doi: 10.1001/jamaneurol.2023.2754. PMID 37603325
- [Derived] Garcia-Tornel A, Flores A, Terceno M, Cardona P, Amaro S, Gomis M, Zaragoza J, Krupinski J, Gomez-Choco M, Mas N, Cocho D, Catena E, Purroy F, Deck M, Rubiera M, Pagola J, Rodriguez-Luna D, Juega J, Rodriguez-Villatoro N, Molina CA, Soro C, Jimenez X, Salvat-Plana M, Davalos A, Jovin TG, Abilleira S, Perez de la Ossa N, Ribo M; RACECAT Trial Investigators. Association of Time of Day With Outcomes Among Patients Triaged for a Suspected Severe Stroke in Nonurban Catalonia. Stroke. 2023 Mar;54(3):770-780. doi: 10.1161/STROKEAHA.122.041013. Epub 2023 Feb 27. PMID 36848432
- [Derived] Garcia-Tornel A, Millan M, Rubiera M, Bustamante A, Requena M, Dorado L, Olive-Gadea M, Jimenez X, Soto A, Querol M, Hernandez-Perez M, Gomis M, Cardona P, Urra X, Purroy F, Silva Y, Ustrell X, Esteve P, Salvat-Plana M, Gallofre M, Molina C, Davalos A, Jovin T, Abilleira S, Ribo M, Perez de la Ossa N; RACECAT Trial Investigators. Workflows and Outcomes in Patients With Suspected Large Vessel Occlusion Stroke Triaged in Urban and Nonurban Areas. Stroke. 2022 Dec;53(12):3728-3740. doi: 10.1161/STROKEAHA.122.040768. Epub 2022 Oct 19. PMID 36259411
- [Derived] Garcia-Tornel A, Sero L, Urra X, Cardona P, Zaragoza J, Krupinski J, Gomez-Choco M, Sala NM, Catena E, Palomeras E, Serena J, Hernandez-Perez M, Boned S, Olive-Gadea M, Requena M, Muchada M, Tomasello A, Molina CA, Salvat-Plana M, Escudero M, Jimenez X, Davalos A, Jovin TG, Purroy F, Abilleira S, Ribo M, de la Ossa NP; RACECAT trial investigators. Workflow Times and Outcomes in Patients Triaged for a Suspected Severe Stroke. Ann Neurol. 2022 Dec;92(6):931-942. doi: 10.1002/ana.26489. Epub 2022 Sep 7. PMID 36053966
- [Derived] Perez de la Ossa N, Abilleira S, Jovin TG, Garcia-Tornel A, Jimenez X, Urra X, Cardona P, Cocho D, Purroy F, Serena J, San Roman Manzanera L, Vivanco-Hidalgo RM, Salvat-Plana M, Chamorro A, Gallofre M, Molina CA, Cobo E, Davalos A, Ribo M; RACECAT Trial Investigators. Effect of Direct Transportation to Thrombectomy-Capable Center vs Local Stroke Center on Neurological Outcomes in Patients With Suspected Large-Vessel Occlusion Stroke in Nonurban Areas: The RACECAT Randomized Clinical Trial. JAMA. 2022 May 10;327(18):1782-1794. doi: 10.1001/jama.2022.4404. PMID 35510397
- [Derived] Abilleira S, Perez de la Ossa N, Jimenez X, Cardona P, Cocho D, Purroy F, Serena J, Roman LS, Urra X, Vilaro M, Cortes J, Gonzalez JA, Chamorro A, Gallofre M, Jovin T, Molina C, Cobo E, Davalos A, Ribo M. Transfer to the Local Stroke Center versus Direct Transfer to Endovascular Center of Acute Stroke Patients with Suspected Large Vessel Occlusion in the Catalan Territory (RACECAT): Study protocol of a cluster randomized within a cohort trial. Int J Stroke. 2019 Oct;14(7):734-744. doi: 10.1177/1747493019852176. Epub 2019 May 29. PMID 31142219